CLINICAL TRIAL: NCT04479995
Title: Multidisciplinary Intervention to Promote Medical Adherence and Coping in Patients With Moderate to Severe Chronic Graft-Versus-Host Disease (GVHD
Brief Title: Multidisciplinary Intervention In Chronic GVHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-772
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stem Cell Transplant Complications; Graft Vs Host Disease; Coping Skills; Quality of Life
Keywords: Stem Cell Transplant Complications; Graft Vs Host Disease; Coping Skills; Quality of Life
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizon Program (Experimental): Eight weekly, audio recorded telehealth videoconferencing sessions. Sessions are 90 minutes.
  Questionnaire assessments at 8 and 16 weeks after end of videoconferencing sessions
  Interventions: Behavioral: Horizon Program
- Usual Care (Experimental): Standard medical visits to address chronic GVHD, with an additional standardized booklet, in electronic or paper format, containing information on the management of chronic GVHD and stem cell transplant survivorship recommendations.
  Questionnaire assessment at 8 weeks and 16 weeks after Horizons Program group starts
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Horizon Program — Telehealth videoconferencing sessions and questionnaires.
  Arms: Horizon Program
Behavioral: Usual Care — Standard medical visits with additional paper or electronic booklet.
  Arms: Usual Care

SUMMARY:
This research is being done to evaluate the feasibility and efficacy of a multidisciplinary, patient-centered intervention, Horizons Program, versus minimally enhanced standard care to improve quality of life, symptom burden and psychological distress of adults who received an allogeneic hematopoietic stem cell transplant and developed graft versus-host disease (GVHD).

DETAILED DESCRIPTION:
This randomized research study is being conducted to see if the Horizons Program compared to usual care is manageable and effective at improving understanding of chronic GVHD and treatment, coping, and quality of life.

Randomization means that participants will be put into one of two groups by chance:

* Horizons Program

  --Individuals who receive the Horizons Program will attend 8 weekly 90-minute group sessions using a secure TeleHealth videoconferencing system
* Usual care --Individuals who receive usual care will also receive an educational booklet.

The research study procedures include:

* screening for eligibility
* a brief test of videoconferencing software
* completion of three study assessments (after signing consent but before randomization and at 8 weeks and 16 weeks after the start of the Horizons Program)
* Individuals who receive usual care will also receive an educational booklet. It is anticipated 80 people will take part in this research study.

The MGH BMT Survivorship Program is supporting this research study by providing funding for this project.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 21 years) who underwent allogeneic HCT
* have moderate to severe chronic GVHD
* are currently receiving their care at the MGH Blood and Marrow Transplant Clinic
* have the ability to participate in an English language group intervention

Exclusion Criteria:

* Patients with comorbid conditions or cognitive impairment that the treating clinician believes prohibits informed consent or participation in the intervention
* Vulnerable patients, defined here as prisoners and pregnant women, will not be included in the intervention

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-02 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Enrollment | Baseline (pre-randomization) to 8 week follow up
  Feasibility will be demonstrated if ≥50% eligible participants enroll
Rate of adherence | Baseline (pre-randomization) to 8 week follow up
  Feasibility will be demonstrated if 80% complete ≥4 of 8 sessions
Rate of retention | Baseline (pre-randomization) to 8 week follow up
  Feasibility will be demonstrated if 80% of participants remain in study

SECONDARY OUTCOMES:
Quality of life (QOL): Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) | Baseline (pre-randomization) up to 16 week follow up
  We will use linear mixed models to investigate longitudinal differences in quality of life between study groups (FACT-BMT score range 0-164, with higher scores indicating better quality of life).
Symptom Burden: Lee Chronic Graft-Versus-Host Disease Symptom Scale (Lee cGVHD) | Baseline (pre-randomization) up to 16 week follow up
  We will use linear mixed models to investigate longitudinal differences in symptom burden between study groups (Lee cGVHD score range 0-56, with higher scores indicating worse symptom burden).
Psychological Distress: Hospital Anxiety and Depression Scale (HADS) | Baseline (pre-randomization) up to 16 week follow up
  We will use linear mixed models to investigate longitudinal differences in psychological distress between study groups (HADS score range 0-21, with higher scores indicating greater distress).
Medical Adherence: Medication Adherence Report Scale (MARS-5) | Baseline (pre-randomization) up to 16 week follow up
  We will use linear mixed models to investigate longitudinal differences in medical adherence self management between study groups (MARS-5 score range 5-25, with higher scores indicating greater adherence).
Social Support: Medical Outcomes Study Social Support Survey (MOS SSS) | Baseline (pre-randomization) up to 16 week follow up
  We will use linear mixed models to investigate longitudinal differences in social support self management between study groups (MOS SSS score range 0-100, with higher scores indicating greater support).
Self-Efficacy: Cancer Self-Efficacy Scale (CASE) | Baseline (pre-randomization) up to 16 week follow up
  We will use linear mixed models to investigate longitudinal differences in cancer self-efficacy between study groups (CASE score range 0-170, with higher scores indicating greater self-efficacy).
Coping Skills: Measure of Current Status (MOCS) | Baseline (pre-randomization) up to 16 week follow up
  Using to compare Coping Skills self management target between study groups
  We will use linear mixed models to investigate longitudinal differences in coping skills between study groups (CASE score range 0-52, with higher scores indicating greater coping skill).

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Centracchio JA, Yang DG, Jagielo AD, Greer JA, El-Jawahri A, Traeger L, Nelson AM. "They knew the same struggles": perceptions of a group coping skills intervention in patients with chronic graft-versus-host disease. Support Care Cancer. 2025 Jan 16;33(2):102. doi: 10.1007/s00520-025-09153-x. PMID 39814942